CLINICAL TRIAL: NCT02537171
Title: Apatinib as Maintenance Therapy After First Line Treatment in Locally Advanced or Metastatic Gastric Cancer: A Randomized, Parallel, Controlled Study
Brief Title: Apatinib as Maintenance Therapy After First Line Treatment in Locally Advanced or Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-G303
Record Dates: First submitted 2015-07-13; First posted 2015-09-01 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2015-08

CONDITIONS: Gastric Cancer
Keywords: Apatinib; Locally Advanced Gastric Cancer; Metastatic Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apatinib 750mg group (Active Comparator): Apatinib mesylate tablets(ATAN) is taken 750mg every day orally, half hour after breakfast with warm water. The drug is taken 4 weeks one cycle until disease progression or intolerable toxicity or death.The dose of the study drug may be modified following the occurence of a clinically significant adverse event(AE).
  Interventions: Drug: apatinib
- Apatinib 500mg group (Active Comparator): Apatinib Mesylate Tablets(ATAN) is taken 500mg every day orally, half hour after breakfast with warm water. The drug is taken 4 weeks one cycle until disease progression or intolerable toxicity or death.Treatment will be discontinued if the subject is unable to tolerate a daily dose of 500mg.
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — Patients will be randomly assigned on a 1:1 basis to treatment with Apatinib 750mg group or Apatinib 500mg group.
  Other Names: ATAN

SUMMARY:
The study is to evaluate the efficacy of Apatinib in patients with advanced or metastatic adenocarcinoma of stomach or gastroesophageal junction.

DETAILED DESCRIPTION:
The study is to investigate the efficacy of Apatinib as maintenance therapy after first fine treatment in patients with advanced or metastatic adenocarcinoma of stomach or gastroesophageal junction through progression-free survival(PFS). Apatinib will be given to patients who have received first-line chemotherapy with an efficacy assessment of stable disease(SD), complete response(CR), or partial response(PR) after 4 cycles. Patients were randomly assigned to 750mg group or 500mg group continually until disease progression or intolerable toxicity or patients withdrawal of consent, and the sample size is 40 individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years;
2. Pathologically diagnosed with advanced gastric adenocarcinoma (including gastroesophageal junction) with measurable metastases outside the stomach (≥10mm on spiral CT scan, and meet the criteria of Response Evaluation Criteria in Solid Tumors 1.1);
3. Locally advanced, recurrent or metastatic gastric or gastro-oesophageal junction adenocarcinoma;
4. Finished first-line chemotherapy (fluorouracil combined with oxaliplatin, cisplatin, paclitaxel or docetaxel) 3 weeks a cycle for 4 cycles, of which the last efficacy assessment is SD, PR or CR. No more than 28 days from the starting day of last cycle of chemotherapy;
5. Eastern Cooperative Oncology Group（ECOG）performance status 0 or 1;
6. Blood routine test and Biochemical tests:

   * Hemoglobin ≥ 80g / L;
   * Absolute neutrophil count (ANC) ≥ 1.5 × 109 / L;
   * Platelet count≥ 90 × 109 / L;
   * Alanine aminotransferase (ALT)and Aspartate aminotransferase (AST) <2.5× upper limit of normal (ULN); liver metastases, if any, the ALT and AST<5 × ULN;
   * Serum total bilirubin≤1.5 × ULN;
   * Serum creatinine≤1.5 × ULN;
   * Serum albumin≥30g/L;
7. Life expectancy more than 3 months;
8. Voluntarily join the study and sign the Informed Consent Form for the study;
9. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. They shall take appropriate methods for contraception during the study until the 8th week post the last administration of study drug. For men, (previous surgical sterilization accepted), shall agree to take appropriate methods of contraception during the study until the 8th week post the last administration of study drug.

Exclusion Criteria:

1. Patients with a known history of allergic reactions and/or hypersensitivity attributed to apatinib or its accessories;
2. Subjects with poor-controlled arterial hypertension (systolic blood pressure> 140 mmHg and diastolic blood pressure > 90 mm Hg) despite standard medical management; Coronary heart disease greater than ClassⅠ; Ⅰ-level arrhythmia (including QT interval prolongation, for man ≥ 450 ms, for woman ≥ 470 ms) together with Class Ⅰcardiac dysfunction; Patients with positive urinary protein;
3. Factors that could have an effect on oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
4. Subjects with high gastrointestinal bleeding risk, including the following conditions: local active ulcer lesions with positive fecal occult blood test (++); history of black stool, or haematemesis in the past 2 months;primary lesion in stomach with positive fecal occult blood test (+) should be evaluated by endoscopy and other potential massive haemorrhage conditions evaluated by the investigator;
5. Abnormal Coagulation (international normalized ratio>1.5, activated partial thromboplastin time>1.5 UNL), with tendency of bleeding;
6. Associated with central nervous system (CNS) metastases;
7. Pregnant or lactating women;
8. Suffering from other malignancies within 5 years;
9. History of uncontrolled psychotropic drug abuse or mental disorders;
10. Participated in other clinical study within 4 weeks;
11. Prior VEGFR inhibitor treatment,such as sorafenib and sunitinib ;
12. Concomitant disease conditions judged by investigator that may seriously affect subject's safety or affect the study completion;
13. Other cases that the researcher found ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
disease control rate(DCR） | 1year
  Investigators will assess treatment response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）
Objective tumor response rate(ORR) | 1year
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
overall survival(OS) | 3year
  OS is defined as the length of time from random assignment to death or to last contact.
Quality of life score （QoL） | 1year
  QoL is a questionnaire developed to assess the quality of life of cancer patients.
Adverse Events(AEs) | 1year
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xu jianming, M.D., Principal Investigator — 307 Hospital of PLA
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China